CLINICAL TRIAL: NCT00127530
Title: Double-Blind, Placebo-Controlled, 21-Week, Parallel Group Study to Evaluate Safety and Efficacy of Oral Fampridine-SR in Subjects With Multiple Sclerosis
Brief Title: Study of Oral Fampridine-SR in Multiple Sclerosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Acorda Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MS-F203
Record Dates: First submitted 2005-08-04; First posted 2005-08-08 (Estimated); Results first posted 2011-05-06 (Estimated); Last update posted 2018-09-11 (Actual); Status verified 2018-08

CONDITIONS: Multiple Sclerosis
Keywords: Walking Ability
MeSH Terms: conditions — Multiple Sclerosis | interventions — 4-Aminopyridine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo- sugar pill (Placebo Comparator): Placebo control
  Interventions: Drug: Placebo
- Fampridine-SR (Experimental): 10 milligram (mg) tablet b.i.d.
  Interventions: Drug: Fampridine-SR

INTERVENTIONS:
Drug: Fampridine-SR — Tablets, 10 mg, twice daily, 14 weeks
  Other Names: Sustained release 4-aminopyridine, 4-AP
  Arms: Fampridine-SR
Drug: Placebo — sugar pill, twice a day (b.i.d.)
  Arms: Placebo- sugar pill

SUMMARY:
To assess the safety and efficacy of 10 milligram (mg) twice a day (b.i.d.) Fampridine-SR in patients diagnosed with multiple sclerosis (MS), in a double-blind, placebo-controlled, parallel group study.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a disorder of the body's immune system that affects the central nervous system (CNS). Normally, nerve fibers carry electrical impulses through the spinal cord, providing communication between the brain and the arms and legs. In people with MS, the fatty sheath that surrounds and insulates the nerve fibers (called "myelin") deteriorates, causing nerve impulses to be slowed or stopped. As a result, patients with MS may experience periods of muscle weakness and other symptoms such as numbness, loss of vision, loss of coordination, paralysis, spasticity, mental and physical fatigue and a decrease in the ability to think and/or remember. These periods of illness may come (exacerbations) and go (remissions). Fampridine-SR is an experimental drug that has been reported to possibly improve muscle strength and walking ability for some people with MS. This study will evaluate the effects and possible risks of taking Fampridine-SR in subjects with MS.

ELIGIBILITY:
Inclusion Criteria:

* Have a confirmed diagnosis of multiple sclerosis
* Are able to walk with or without an assistive device

Exclusion Criteria:

* Pregnancy, breastfeeding or females of childbearing potential not using adequate birth control
* Participating in other investigational drug trials
* A medical history or clinical findings that preclude entry into the study
* A medication history that precludes entry into the study
* Previously treated with 4-aminopyridine (4-AP)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2005-05; Primary Completion 2006-06 (Actual); Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Blight, PhD, Study Director — Acorda Therapeutics
Locations (34):
- United States (30):
  - University of Alabama, Birmingham, Alabama
  - Barrow Neurology Clinic, St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - USC, Keck School of Medicine, Los Angeles, California
  - UC Davis, Sacramento, California
  - University of Colorado Health Sciences Center, Denver, Colorado
  - Multiple Sclerosis Treatment Center, Derby, Connecticut
  - Shepard Center, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Indiana University MS Center, Indianapolis, Indiana
  - Maryland Center for MS, Baltimore, Maryland
  - Wayne State University, Department of Neurology, Detroit, Michigan
  - The Schapiro Center for MS, Golden Valley, Minnesota
  - Washington University SOM, St Louis, Missouri
  - Gimbel MS Center at Holy Name Hospital, Teaneck, New Jersey
  - University of Mexico, MIND Imaging Center, Albuquerque, New Mexico
  - Maimonides Medical Center, Brooklyn, New York
  - Corinne Goldsmith Dickinson Center for MS, New York, New York
  - University of Rochester, Rochester, New York
  - SUNY - Stony Brook, Stony Brook, New York
  - Carolinas Healthcare System, Charlotte, North Carolina
  - Cleveland Clinical Foundation, Cleveland, Ohio
  - Ohio State University MS Center, Columbus, Ohio
  - Oregon Health & Science University, MS Center of Oregon, UHS-42, Portland, Oregon
  - Thomas Jefferson University Physicians, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Allegheny Neurological Associates, Pittsburgh, Pennsylvania
  - University of Texas - Houston, Houston, Texas
  - Neurological Research Center, Inc., Bennington, Vermont
  - Fletcher Allen Health Care, Burlington, Vermont
  - MS Hub Medical Group, Seattle, Washington
  - University of Washington, MS Research Center, Seattle, Washington
- Canada (4):
  - Foothills Medical Center, Calgary, Alberta
  - University of British Columbia, Vancouver Coastal Health Research Institute, Vancouver, British Columbia
  - QEII Health Sciences Centre, Nova Scotia Rehabilitation Centre Site, Halifax, Nova Scotia
  - Ottawa Hospital General Campus, Ottawa, Ontario

REFERENCES:
- [Result] Goodman AD, Brown TR, Krupp LB, Schapiro RT, Schwid SR, Cohen R, Marinucci LN, Blight AR; Fampridine MS-F203 Investigators. Sustained-release oral fampridine in multiple sclerosis: a randomised, double-blind, controlled trial. Lancet. 2009 Feb 28;373(9665):732-8. doi: 10.1016/S0140-6736(09)60442-6. PMID 19249634

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo- Sugar Pill: Placebo control group
- Fampridine-SR: 10 milligram (mg) tablet twice a day (b.i.d.)
Period: Overall Study
Arm/Group | Placebo- Sugar Pill | Fampridine-SR
Started | 72 | 228
Completed | 71 | 207
Not Completed | 1 | 21

BASELINE CHARACTERISTICS:
Population: Safety Population = Placebo (72), Fampridine-SR (228) Intent to Treat (ITT) Population = Placebo (72), Fampridine-SR (224).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo- Sugar Pill | Fampridine-SR | Total
Number analyzed (Participants) | 72 | 228 | 300
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.9 (8.88) | 51.5 (8.72) | 51.4 (8.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 162 | 205
  Male | 29 | 66 | 95
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 67 | 211 | 278
  Black | 3 | 10 | 13
  Hispanic | 1 | 3 | 4
  Asian/Pacific Islander | 1 | 3 | 4
  Other | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Timed Walk Responders (Patients Who Showed Consistent Improvement on the Timed-25 Foot Walk)
Description: Patients who showed a faster walking speed for at least three of the four on-drug visits during the double-blind treatment period as compared to the maximum speed for any of the five off-drug visits.
Time Frame: Days 14, 42, 70 and 98 of treatment, corresponding to the four on-drug visits during double-blind treatment period.
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo- Sugar Pill | Fampridine-SR
Number analyzed (Participants) | 72 | 224
Participants | 6 | 78

2. Secondary Outcome: Lower Extremity Manual Muscle Test; Ashworth Score for Spasticity
Time Frame: Days 14, 42, 70, 98
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Placebo- Sugar Pill | Fampridine-SR
Serious Adverse Events (participants affected / at risk) | 0/72 | 16/228
Other Adverse Events (participants affected / at risk) | 58/72 | 191/228
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo- Sugar Pill (N=72) | Fampridine-SR (N=228)
Angina pectoris (Vascular disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Multiple sclerosis (Nervous system disorders) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo- Sugar Pill (N=72) | Fampridine-SR (N=228)
asthenia (Musculoskeletal and connective tissue disorders) | 4 (5) | 13 (16)
back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 13 (14)
balance disorder (Nervous system disorders) | 2 (2) | 13 (13)
dizziness (Nervous system disorders) | 4 (4) | 19 (21)
fall (Injury, poisoning and procedural complications) | 11 (14) | 36 (56)
fatigue (General disorders) | 2 (2) | 14 (15)
headache (Nervous system disorders) | 4 (4) | 13 (14)
insomnia (Nervous system disorders) | 3 (3) | 19 (21)
Nausea (Gastrointestinal disorders) | 3 (3) | 14 (16)
Upper Respiratory Tract infection (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 14 (17)
Urinary Tract Infection (Infections and infestations) | 10 (11) | 31 (40)
Multiple Sclerosis (Vascular disorders) | 2 | 11
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 4 | 10
Paraesthesia (Nervous system disorders) | 4 | 10
Hypoaesthesia (Nervous system disorders) | 4 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor (Acorda) has right to review and comment on proposed publications within a specified time frame, up to 60 days; multi-center trials require joint publication unless specifically permitted otherwise.